CLINICAL TRIAL: NCT02419482
Title: Improving Reproductive Function in Women With Polycystic Ovary Syndrome by High Intensity Interval Training: A Randomized Controlled Trial.
Brief Title: Improving Reproductive Function in Women With Polycystic Ovary Syndrome by High Intensity Interval Training
Acronym: IMPROV-IT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); Liverpool John Moores University (Other); Australian Catholic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015/468
Record Dates: First submitted 2015-04-14; First posted 2015-04-17 (Estimated); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Exercise therapy; Reproductive Physiological Processes; Fertility
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — High-Intensity Interval Training; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 4x4 minutes interval training (Experimental): 4x4 minutes high intensity interval training with 4 minute intervals
  Interventions: Behavioral: 4x4 minutes high intensity interval training
- 10x1 minute interval training (Experimental): 10x1 minute high intensity interval training with 1 minute intervals
  Interventions: Behavioral: 10x1 minute high intensity interval training
- control (No Intervention): Physical activity recommended

INTERVENTIONS:
Behavioral: 4x4 minutes high intensity interval training — Treadmill running/walking with 10 minutes varm-up at 60-70% of maximum heart rate, 4x4 minute intervals at 90-95% of maximum heart rate separated by 3-minutes active pauses at 60-70% of maximum heart rate, and 3 minutes cool-down.
  Other Names: High-intensity exercise; Aerobic exercise
  Arms: 4x4 minutes interval training
Behavioral: 10x1 minute high intensity interval training — Treadmill running/walking with 10 minutes varm-up at 60-70% of maximum heart rate, ten 1-minute intervals at maximal intensity (that can be performed for one minute), separated by 1-minutes active pauses at 60-70% of maximum heart rate, and 3 minutes cool-down.
  Other Names: High-intensity exercise; Aerobic exercise
  Arms: 10x1 minute interval training

SUMMARY:
The aim is to investigate whether 16 weeks of high intensity interval training, followed by 36 weeks of home-based exercise, will improve menstrual frequency in women with Polycystic Ovary Syndrome (PCOS) compared with a non-exercising control group.

ELIGIBILITY:
Inclusion Criteria:

* Polycystic ovary syndrome (PCOS) according to the Rotterdam criteria

Exclusion Criteria:

* Regular high intensity endurance (two or more times per week of vigorous exercise).
* Concurrent treatments (insulin sensitizers or drugs known to affect gonadotropin or ovulation, with a wash out period of 1 months prior to inclusion).
* On-going pregnancy.
* Breast feeding within 24 weeks
* Cardiovascular disease or endocrine disorders

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Menstrual frequency | 1 year
  Electronic menstrual diary

SECONDARY OUTCOMES:
Body composition | 16 weeks, and 36 weeks
  Bioimpedance scale and/or DXA, waist circumference, waist/hip-ratio
Aerobic capacity | 16 weeks, and 36 weeks
  Maximal oxygen uptake measured with Oxygon Pro, Jaeger
Endothelial function | 16 weeks, and 36 weeks
  Flow mediated dilatation of the brachial artery
Insulin sensitivity | 16 weeks, and 36 weeks
  2h oral glucose tolerance test (OGGT)
Intima-media thickness | 16 weeks, and 36 weeks
  Ultrasound of the caroid intima-media thickness
Oxidative capacity | 16 weeks, and 36 weeks
  carbohydrate- and fat oxidation measured with Oxygon Pro, Jaeger
Low-grade systematic inflammation | 16 weeks, and 36 weeks
  Blood samples and adipose tissue
Adipose tissue morphology and function | 16 weeks, (and 36 weeks if funded)
  Adipose tissue biopsy
Hormone profile, blood lipids and blood values | 16 weeks, and 36 weeks
  Blood samples
Blood pressure | 16 weeks, and 36 weeks
  Systolic and diastolic measured with automatic blood pressure device
Quality of life | 16 weeks
  PCOS-specific Quality of Life Questionnaire
Quality of life | 36 weeks
  PCOS-specific Quality of Life Questionnaire
Physical activity | 16 weeks, and 36 weeks
  Physical activity monitor armband (amount and intensity)
Adipose tissue mRNA expression | 16 weeks, (and 36 weeks if funded)
  mRNA analysis of adipose tissue
ovarian morphology | 16 weeks, and 36 weeks
  vaginal ultrasound
Pregnancy rate | 16 weeks , and 36 weeks
  In total, between groups, and among those trying to become pregnant when entering the study
Enjoyment | weekly up to 16 weeks
  Physical Activity Enjoyment Scale (PACES) questionnaire
Diet | 16 weeks
  Diet diary
Diet | 36 weeks
  Diet diary

CONTACTS AND LOCATIONS:
Overall Officials: Trine Moholdt, phd, Principal Investigator — Norwegian University of Science and Technology
Locations (2):
- Centre of Exercise and Nutrition, Mary MacKillop Institute for Health Research, AUC, Melbourne, Australia
- Department of circulation and medical imaging , NTNU, Trondheim, Norway

REFERENCES:
- [Result] Lionett S, Kiel IA, Camera DM, Vanky E, Parr EB, Lydersen S, Hawley JA, Moholdt T. Circulating and Adipose Tissue miRNAs in Women With Polycystic Ovary Syndrome and Responses to High-Intensity Interval Training. Front Physiol. 2020 Jul 30;11:904. doi: 10.3389/fphys.2020.00904. eCollection 2020. PMID 32848854
- [Derived] Kiel IA, Lionett S, Parr EB, Jones H, Roset MAH, Salvesen O, Hawley JA, Vanky E, Moholdt T. High-Intensity Interval Training in Polycystic Ovary Syndrome: A Two-Center, Three-Armed Randomized Controlled Trial. Med Sci Sports Exerc. 2022 May 1;54(5):717-727. doi: 10.1249/MSS.0000000000002849. Epub 2022 Jan 12. PMID 35019901
- [Derived] Lionett S, Kiel IA, Rosbjorgen R, Lydersen S, Larsen S, Moholdt T. Absent Exercise-Induced Improvements in Fat Oxidation in Women With Polycystic Ovary Syndrome After High-Intensity Interval Training. Front Physiol. 2021 Mar 24;12:649794. doi: 10.3389/fphys.2021.649794. eCollection 2021. PMID 33841184
- [Derived] Kiel IA, Lionett S, Parr EB, Jones H, Roset MAH, Salvesen O, Vanky E, Moholdt T. Improving reproductive function in women with polycystic ovary syndrome with high-intensity interval training (IMPROV-IT): study protocol for a two-centre, three-armed randomised controlled trial. BMJ Open. 2020 Feb 20;10(2):e034733. doi: 10.1136/bmjopen-2019-034733. PMID 32086359